CLINICAL TRIAL: NCT07066059
Title: Study on the Efficacy and Safety of Shouhui Tongbian Capsules in Protecting Intestine During the Perioperative Period
Status: Not yet recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Shandong University (Other)
Collaborators: Shandong Public Health Clinical Center (Other Government)
Responsible Party: Principal Investigator, Wei Zhao, Head of department of clinical pharmacy and pharmacology, Shandong University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SDU-2025-XM-002
Record Dates: First submitted 2025-06-25; First posted 2025-07-15 (Actual); Last update posted 2025-07-15 (Actual); Status verified 2025-07

CONDITIONS: Perioperative Period

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard Treatment group (No Intervention): Receive routine perioperative care including diet control and standard bowel-cleansing drugs
- Shouhui Tongbian Capsules group (Experimental): Receive Shouhui Tongbian Capsules
  Interventions: Drug: Shouhui Tongbian Capsules

INTERVENTIONS:
Drug: Shouhui Tongbian Capsules — 2 pills twice daily from admission to the night before surgery, then resuming after bowel sound recovery and oral intake postoperatively, with a 3-day post-discharge regimen
  Arms: Shouhui Tongbian Capsules group

SUMMARY:
The goal of this clinical trial is to investigate if Shouhui Tongbian Capsules can shorten intestinal function recovery time (exhaust/defecation time) and improve defecation quality in perioperative patients, and to evaluate its safety and comfort advantages during the perioperative period. The study involves participants aged 18-70 years, both male and female, with ASA grade I-III scheduled for elective surgery. The main questions it aims to answer are:

Can Shouhui Tongbian Capsules shorten the intestinal function recovery time (first flatus and defecation time) in perioperative patients? Can Shouhui Tongbian Capsules improve defecation quality (assessed by Bristol Stool Scale) and reduce inflammatory factor levels (e.g., IL-6, TNF-α)? Researchers will compare the experimental group (receiving Shouhui Tongbian Capsules 2 pills twice daily from admission to the night before surgery, then resuming after bowel sound recovery and oral intake postoperatively, with a 3-day post-discharge regimen) to the control group (receiving routine perioperative care including diet control and standard bowel-cleansing drugs) to see if the capsules show superior efficacy in intestinal function recovery and safety.

Participants will:

Take Shouhui Tongbian Capsules according to the specified regimen (experimental group) or receive routine care (control group).

Have their exhaust/defecation status recorded every 6 hours postoperatively. Undergo blood tests for liver/kidney function and inflammatory factors on the day before surgery and day 3 postoperatively.

Complete questionnaires on bowel preparation comfort and postoperative defecation satisfaction.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18-70 years, regardless of gender;
2. ASA class I-III, elective surgery patients;
3. Signed the informed consent form.

Exclusion Criteria:

1. Disease-related exclusions:

   Digestive system diseases: intestinal obstruction, intestinal perforation, acute peritonitis; inflammatory bowel disease (ulcerative colitis, Crohn's disease); gastrointestinal tumors (primary or metastatic); severe hemorrhoids or anal fissures (grade Ⅲ-Ⅳ); severe liver disease (Child-Pugh class ≥ B); Other systemic diseases: severe cardiovascular diseases (cardiac function grade Ⅲ or above, severe arrhythmia); uncontrolled diabetes (fasting blood glucose > 11.1 mmol/L); autoimmune diseases (such as active systemic lupus erythematosus, rheumatoid arthritis); advanced malignant tumors or during radiotherapy/chemotherapy.
2. Liver and kidney function abnormalities:

   Alanine aminotransferase (ALT) or aspartate aminotransferase (AST) > 2 times the upper limit of normal (ULN); serum creatinine (Cr) > 1.5 times ULN; estimated glomerular filtration rate (eGFR) < 60 mL/min/1.73 m².
3. Medication-related exclusions:

   Use of the following drugs within the past 2 weeks:

   Laxatives (e.g., lactulose, polyethylene glycol), gastrointestinal motility agents (e.g., domperidone, mosapride), antibiotics (systemic use), opioid analgesics, anticholinergic drugs, long-term laxative use (continuous use ≥ 2 weeks), preoperative use of enteral nutrition preparations or intravenous nutritional support.
4. Exclusions for special populations:

   Pregnant or lactating women; those allergic to components of Shouhui Tongbian Capsules (including Chinese herbal ingredients such as ginseng, atractylodes, polygonum multiflorum); patients with mental disorders or cognitive impairment; emergency or urgent surgery patients; those with an expected postoperative hospital stay < 3 days.
5. Other exclusions:

Participation in other clinical trials without passing the washout period; other situations where the investigator deems the subject unsuitable for the study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2025-08-01 (Estimated); Primary Completion 2027-03-31 (Estimated); Study Completion 2027-07-31 (Estimated)

PRIMARY OUTCOMES:
Postoperative intestinal function recovery time | Throughout the study drug treatment period, about 2 weeks
  Observe and record the postoperative intestinal function recovery time of the two groups of patients (including the time of first exhaust and defecation). The shorter the time, the better.
Total duration of intestinal function recovery | Throughout the study drug treatment period, about 2 weeks
  Observe and record the total duration of intestinal function recovery of the two groups of patients. The shorter the time, the better.
Defecation trait score | Throughout the study drug treatment period, about 2 weeks
  Observe and record the defecation trait score of the two groups of patients (using the Bristol Stool Scale). Seven types of stools based on shape and consistency, with type 1 being the hardest and type 7 being the softest
Levels of inflammatory factors | Throughout the study drug treatment period, about 2 weeks
  Measure the levels of inflammatory factors (such as IL-6, TNF-α, etc.).

SECONDARY OUTCOMES:
Adverse event rate | Throughout the study drug treatment period, about 2 weeks
  Record adverse events occurring in the two groups of patients during the study period, including gastrointestinal discomfort (nausea, vomiting, abdominal pain, etc.), changes in liver and kidney function indicators, etc.
Comfort of intestinal preparation satisfaction questionnaire | Throughout the study drug treatment period, about 2 weeks
  Evaluate the differences in comfort of intestinal preparation satisfaction between the two groups of patients through questionnaires. The higher the score, the better.
Postoperative defecation satisfaction questionnaire | Throughout the study drug treatment period, about 2 weeks
  Evaluate the differences in postoperative defecation satisfaction between the two groups of patients through questionnaires. The higher the score, the better.

CONTACTS AND LOCATIONS:
Overall Officials: Qiang Zhang, Principal Investigator — Shandong Public Health Clinical Center
Locations (1):
- Shandong Public Health Clinical Center, Jinan, China

IPD SHARING:
Plan to Share IPD: Undecided